CLINICAL TRIAL: NCT05412836
Title: Intra-Articular Injection in Moderate Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lipo-Sphere (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJO-01
Record Dates: First submitted 2022-02-27; First posted 2022-06-09 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One Treatment Arm (Experimental): Subjects will receive a single intra-articular injection of AqueousJoint.
  Interventions: Device: AqueousJoint

INTERVENTIONS:
Device: AqueousJoint — AqueousJoint is a liposomal boundary lubricant, which coats the cartilage surface and protects it from further damage and degradation.

SUMMARY:
AqueousJoint is a new intra-articular (IA) injectable joint lubricant for patients suffering from knee Osteoarthritis developed by Liposphere LTD.

AqueousJoint is a liposomal boundary lubricant, which coats the cartilage surface and protects it from further damage and degradation. The product goal is restoring cartilage its natural bio-lubrication properties.

AqueousJoint is a surface lubricant that does not change the synovial fluid mechanical characterization but provides hydration protection from cartilage degradation and wear.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
* Adult male or female at age ≥40 and ≤ 80 years old
* Pain in the intended study knee with an average VAS score of >5 over the last week prior to visit 1 (pre-injection).
* Degenerative changes in the intended study knee that can be categorized as grade II-IV Kellgren Lawrence based upon standing posterior-anterior and lateral radiographs of the knee based on X-RAY from up to the last 6 months prior visit 1 (pre-injection).
* Body Mass Index (BMI) between 18.5 and 35.
* A negative urine pregnancy test female patient with childbearing potential at Visit 1 prior to intra-articular injection of AqueousJoint.
* If female, subject must be either postmenopausal, OR permanently surgically sterile OR for women of childbearing potential using at least 2 methods of birth control that are effective from at least 30 days before Visit 1 through visit 26w (26 weeks post injection).
* Are willing or able to comply with procedures required in this protocol.

Exclusion Criteria:

* History of significant knee trauma or previous arthroscopic surgery of the intended study knee within the last 3 months preceding screening.
* Concomitant moderate or large size synovial fluid effusion of the index knee at Screening
* Wound in the area of the intended study knee
* Fever signs or symptoms of systemic infection or infection of the intended study knee, on the day before or the day of administration of treatment.
* Intra-articular injection to the intended study knee within 3 months prior to Screening.
* Intra-articular injection was administrated during the past 6 weeks
* Intake of chronic pain medications (especially opioid pain relievers) without an option to pause for the period of the study
* Pain in any other joints with an average VAS score (active) of >4 at the time of Visit 1.
* History of Psoriatic Arthritis, Rheumatoid Arthritis or any other inflammatory condition associated with arthritis
* Known history of a severe allergic reaction
* Known Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS), Known Hepatitis B or C viral
* history of clinically significant renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, pulmonary or hepatic disease within the last 6 months that, in the Investigator's opinion, would adversely affect the subject's participation in the study.
* History of cellulitis of the lower extremities, a peripheral vascular disease.
* History of malignancies during the pat 3 years
* Life expectancy of less than 12 month
* Surgery involving the chest, abdomen, pelvis, or lower extremities in the past year
* Participate in other clinical trials within 3 months prior to the study or concurrent with the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events will be evaluated in order to assess the safety of intra-articular injection of Aqueous Joint in osteoarthritic patients up to 26 weeks of follow-up in an open-label clinical study. | 26 weeks
  The safety parameters will include adverse reactions related to the injected material; injection-related side effects consisted of injection-site reaction, erythema, swelling, injection-site pain, and pruritus.

SECONDARY OUTCOMES:
Change in range of motion from visit 1 (pre-injection) to week 26 | 26 weeks
  To measure the effectiveness of the treatment on a range of motion by physical examination
Change in life quality from visit 1 (pre-injection) to week 26 | 26 weeks
  To measure the effectiveness of the treatment on life quality by SF12 Questionnaire
Change in functionality from visit 1 (pre-injection) to week 26 | 26 weeks
  To measure the effectiveness of the treatment on functionality using PRO: KOOS and Physical activity test - Timed up and go examination
Change in pain level and analgesics consumption from visit 1 (pre-injection) to week 26 | 26 weeks
  To measure the effectiveness of the treatment on pain level using VAS and concomitant medication log

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No